CLINICAL TRIAL: NCT04756804
Title: A Randomized, Controlled Clinical Trial Evaluating A Novel Perioperative Patient Skin Antiseptic Preparation
Brief Title: Perioperative Patient Skin Antiseptic Preparation Evaluation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zurex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZXZP0113
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 70% Isopropyl Alcohol novel preoperative skin antiseptic (Experimental): 70% v/v Isopropyl Alcohol novel preoperative skin antisepsis preparation
  Interventions: Drug: 70% v/v Isopropyl Alcohol Surgical Solution
- 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol preoperative skin antiseptic (Active Comparator): 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol preoperative skin antisepsis preparation
  Interventions: Drug: 2%w/v Chlorhexidine Gluconate / 70% v/v Isopropyl Alcohol

INTERVENTIONS:
Drug: 70% v/v Isopropyl Alcohol Surgical Solution — Patient preoperative skin preparation
  Other Names: ZuraGard
  Arms: 70% Isopropyl Alcohol novel preoperative skin antiseptic
Drug: 2%w/v Chlorhexidine Gluconate / 70% v/v Isopropyl Alcohol — Patient preoperative skin preparation
  Other Names: ChloraPrep
  Arms: 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol preoperative skin antiseptic

SUMMARY:
This study will evaluate a new topical skin antiseptic perioperative preparation and the standard of care to determine efficacy on the rates of surgical site infections of surgical patients. Safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female and at least 18 years of age.
2. Be able to verbalize an understanding of the consent form, able to provide written informed consent, verbalize willingness to complete study procedures, able to understand written and oral instructions in English.
3. Be planning to undergo clean (class I wound) or clean-contaminated (class II wounds) surgery.
4. Expect to be available for up to 30-days after the surgery.

Exclusion Criteria:

1. Active infection or fever including evidence of infection at or adjacent to the operative site.
2. Immunosuppressed.
3. Kidney/liver failure.
4. Immunosuppressive therapy (chemotherapy, steroids) within the previous 1 week.
5. Any history of allergy to chlorhexidine or isopropyl alcohol or any other component in ZuraGard including citric acid, sodium citrate, methylparaben, or propylparaben, and FD&C Yellow #6.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Hart, MD, FACS, DFSVS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- MCW/FH, Milwaukee, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 70% Isopropyl Alcohol Novel Preoperative Skin Antiseptic | 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol Preoperative Skin Antiseptic
Started | 25 | 26
Completed | 25 | 25
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 70% Isopropyl Alcohol Novel Preoperative Skin Antiseptic | 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol Preoperative Skin Antiseptic | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 14 | 15 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 10 | 15 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Surgical Site Infection Occurrence
Description: The primary objective is to demonstrate efficacy in surgical use through the rate of surgical site infections.
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 70% Isopropyl Alcohol Novel Preoperative Skin Antiseptic | 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol Preoperative Skin Antiseptic
Number analyzed (Participants) | 25 | 26
Participants | 0 | 1
Statistical Analysis 1: Comparison: 70% Isopropyl Alcohol Novel Preoperative Skin Antiseptic vs 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol Preoperative Skin Antiseptic; Test type: Other — This was a descriptive study, no hypothesis testing was performed; This was a descriptive study, no hypothesis testing was performed

2. Primary Outcome: Allergic Reaction and Skin Irritation
Description: The primary safety objective is to determine the rates of skin irritation or allergic reactions attributed to each drug product and all other adverse events.
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 70% Isopropyl Alcohol Novel Preoperative Skin Antiseptic | 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol Preoperative Skin Antiseptic
Number analyzed (Participants) | 25 | 26
Participants | 1 | 1

3. Secondary Outcome: Subgroup Analysis of Rates of Surgical Site Infections
Description: Surgical site infection rates by different infection types classified as superficial incisional infection, deep incisional infection, or organ-space infection.
Time Frame: Within 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 70% Isopropyl Alcohol Novel Preoperative Skin Antiseptic | 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol Preoperative Skin Antiseptic
Number analyzed (Participants) | 25 | 26
Participants
  superficial incisional infection | 0 | 0
  deep incisional infection | 0 | 1
  organ-space infection | 0 | 0
  No surgical site infection present | 25 | 25

4. Secondary Outcome: Subgroup Analysis of Rates of Surgical Site Infections
Description: Surgical site infection rates by type of surgery including clean (class I wound) or clean-contaminated (class II wounds) surgeries
Time Frame: Within 30 days after surgery
Population: Secondary outcome categorizes the results of the primary outcome - surgical site infections. The study only resulted in observation of 1 surgical site infection in one of the two interventions. Therefore, the novel prep secondary outcome results in a zero value reported.
Measure: Count of Participants; unit: Participants
Arm/Group | 70% Isopropyl Alcohol Novel Preoperative Skin Antiseptic | 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol Preoperative Skin Antiseptic
Number analyzed (Participants) | 0 | 1
Participants
  Class I - Clean | 0 | 1
  Class II - Clean-Contaminated | 0 | 0

ADVERSE EVENTS:
Time Frame: AE's reported from time of enrollment through follow up (30 days post op), up to 51 days ( up to 21 days for screening).
Arm/Group | 70% Isopropyl Alcohol Novel Preoperative Skin Antiseptic | 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol Preoperative Skin Antiseptic
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/26
Serious Adverse Events (participants affected / at risk) | 10/25 | 11/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 70% Isopropyl Alcohol Novel Preoperative Skin Antiseptic (N=25) | 2% Chlorhexidine Gluconate/70% Isopropyl Alcohol Preoperative Skin Antiseptic (N=26)
Cardiac Distress (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal Distress (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Blood Loss Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Heart Failure Exacerbation (Cardiac disorders) | 1 (1) | 1 (1)
Lactic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Outcome fatal, 2 days post op.
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Outcome fatal, 2 days post op.
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1) — Outcome fatal, 2 days post op.
Acute Circulatory Failure (Vascular disorders) | 0 (0) | 1 (1) — Outcome fatal, 2 days post op.
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1) — Outcome fatal, 2 days post op.
Occlusion of Renal Artery (Renal and urinary disorders) | 0 (0) | 1 (1)
Cerebral Hyperperfusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Hypervolemic Shock (Vascular disorders) | 0 (0) | 1 (1)
Altered Mental State (Psychiatric disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Endoleak (General disorders) | 1 (1) | 0 (0)
TIA (Nervous system disorders) | 0 (0) | 1 (1)
Surgical Site Infection (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a pilot study of surgical patients, the majority of which had significant comorbidities with several AEs reported in more than one patient across the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT04756804/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT04756804/SAP_001.pdf